CLINICAL TRIAL: NCT03631043
Title: A Personalized Vaccine for the Immune Prevention of Multiple Myeloma
Brief Title: Personalized Vaccine in Treating Patients With Smoldering Multiple Myeloma
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0345; NCI-2018-01614 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0345 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2018-08-10; First posted 2018-08-15 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Smoldering Plasma Cell Myeloma
MeSH Terms: conditions — Smoldering Multiple Myeloma | interventions — Lenalidomide; Immunotherapy, Active

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Stage I (personalized vaccine) (Experimental): Patients undergo collection of blood and bone marrow for making the vaccine. Patients then receive personalized vaccine SC on days 1 and 15 of cycles 1-2 and on day 1 of cycles 3-6. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Biopsy Specimen Radiography; Biological: Vaccine Therapy
- Stage II (personalized vaccine, lenalidomide) (Experimental): Patients undergo collection of blood and bone marrow for making the vaccine. Patients then receive personalized vaccine SC on days 1 and 15 of cycles 1-2 and on day 1 of cycles 3-6. Patients also receive lenalidomide PO on days 1-21. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Biopsy Specimen Radiography; Drug: Lenalidomide; Biological: Vaccine Therapy

INTERVENTIONS:
Procedure: Biopsy Specimen Radiography — Undergo collection of blood and bone marrow
  Other Names: Biospecimen Radiography; Specimen Radiography
Drug: Lenalidomide — Given PO
  Other Names: CC-5013; CC5013; CDC 501; Revlimid
  Arms: Stage II (personalized vaccine, lenalidomide)
Biological: Vaccine Therapy — Given personalized vaccine SC

SUMMARY:
This early phase I trial studies the side effects of personalized vaccine in treating patients with smoldering multiple myeloma. Vaccines made from a person's blood and bone marrow may help the body build an effective immune response to kill cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To demonstrate that developing a custom vaccine for smoldering multiple myeloma (SMM) is feasible.

II. To show that a custom peptide-based vaccine in smoldering multiple myeloma is safe.

SECONDARY OBJECTIVES:

I. To determine the intensity and longevity of antigen specific T-cell mediated immune responses to the neoantigen vaccine.

II. Time to progression to multiple myeloma (TTM) at the end of the follow up period (18 months).

III. Duration of response. IV. Clinical benefit rate (minor response [MR] or better) after 6 cycles of vaccine treatment per modified International Myeloma Working Group (IMWG) criteria for multiple myeloma (MM).

V. Overall survival.

EXPLORATORY OBJECTIVES:

I. Rate of minimal residual disease (MRD) negativity at complete remission (CR), if achieved. MRD assessment will be based on bone marrow aspirates.

II. Molecular profiling (including whole exome sequencing, gene expression profiling and ribonucleic acid (RNA) sequencing of tumor/bone marrow samples) and cellular (including flow cytometry) profiling at baseline using bone marrow aspirate samples and peripheral blood.

III. Immunophenotypic characterization of dendritic, T-, B-, natural killer (NK)- and NKT-cells, and inhibitory/activation markers on tumor cells at baseline (bone marrow and peripheral blood), day 1 of each cycle (peripheral blood only) and at completion of 6 cycles of therapy (bone marrow and peripheral blood) in bone marrow aspirate samples and/or peripheral blood.

IV. Perform mass spectrometry-based proteomics analysis on 15 myeloma cell lines to identify shared human leukocyte antigen (HLA) class I-restricted antigens that can be targeted with immunotherapy.

OUTLINE: Patients are assigned to 1 of 2 stages.

STAGE I: Patients undergo collection of blood and bone marrow for making the vaccine. Patients then receive personalized vaccine subcutaneously (SC) on days 1 and 15 of cycles 1-2 and on day 1 of cycles 3-6. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.

STAGE II: Patients undergo collection of blood and bone marrow for making the vaccine. Patients then receive personalized vaccine SC on days 1 and 15 of cycles 1-2 and on day 1 of cycles 3-6. Patients also receive lenalidomide orally (PO) on days 1-21. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with intermediate or high-risk smoldering multiple myeloma (SMM) are eligible
* Patients must have histologically confirmed SMM based on the following criteria. Both criteria must be met: (a) Serum monoclonal protein (IgG or IgA) >= 3 g/dL or urinary monoclonal protein >=500 mg per 24 hours and/or clonal bone marrow plasma cells more or equal to 10% (b) Absence of myeloma defining events or amyloidosis
* Additionally, patients must meet criteria for intermediate or high risk of progression to multiple myeloma by Programa para el Estudio de la Terapeutica en Hemopatía Maligna (PETHEMA) criteria (patients must have at least 1 risk factors present):

  * >= 95% abnormal plasma cells/total plasma cells in bone marrow compartment. (This is measured as a percentage of the total abnormal versus normal plasma cells in the bone marrow compartment using standard flow cytometry of the bone marrow aspirate. Having >= 95% abnormal plasma cells/total plasma cells constitutes a risk factor for progression to multiple myeloma by PETHEMA criteria)
  * Immunoparesis (The patient having low uninvolved immunoglobulins in peripheral blood, for example if a patient has IgA smoldering multiple myeloma, then either having a low IgM and/or low IgG will qualify as a risk factor for progression to multiple myeloma) *1 of 2 risk factors: intermediate risk for progression at a rate of ~50% at 5 years *2 of 2 risk factors: high risk for progression at a rate of 72% at 5 years
* Creatinine clearance >= 40 ml/min using the modification of diet in renal disease (MDRD) equation
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Absolute neutrophil count (ANC) >= 1.0 x 10^9/L
* Hemoglobin >= 10 g/dL
* Platelet count >= 50 x 10^9/L
* Platelet and blood transfusions are allowed on protocol. Growth factors, including granulocyte colony stimulating factors and erythropoietin are allowed
* Bilirubin < 1.5 x the upper limit of normal (ULN)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 3.0 x ULN
* Subjects must be able to give informed consent

Exclusion Criteria:

* Evidence of myeloma defining events due to underlying plasma cell proliferative disorder meeting at least one of the following

  * Hypercalcemia: serum calcium > 0.25 mmol/L (> 1 mg/dL) higher than the upper limit of normal or > 2.75 mmol/L (> 11 mg/dL)
  * Renal Insufficiency: creatinine clearance < 40 ml/min or serum creatinine > 2 mg/dL
  * Anemia: hemoglobin value < 10 g/dL
  * Bone lesions: one or more osteolytic lesions on skeletal radiography, computerized tomography (CT) or 2-deoxy-2[F-18] fluoro-D-glucose positron emission tomography CT (PET-CT)
* Prior or concurrent systemic treatment for SMM

  * Bisphosphonates are permitted
  * Treatment with corticosteroids is not permitted (allowed for physiologic doses)
  * Radiotherapy is not permitted
  * Prior treatment for smoldering multiple myeloma with chemotherapy agents approved for the treatment of multiple myeloma is not permitted
* Plasma cell leukemia
* Pregnant or lactating females
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment
* Has a known history of active TB (Bacillus tuberculosis)
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer
* Has an active infection requiring systemic therapy
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 60 days after the last dose of trial treatment
* Has a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies)
* Has known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-12-21 (Actual); Primary Completion 2025-12-10 (Actual); Study Completion 2025-12-10 (Actual)

PRIMARY OUTCOMES:
Feasibility assessed by the proportion of participants for whom the vaccine is successfully developed and ready to administer | Within 12 weeks
Incidence of adverse events | Up to 12 months

SECONDARY OUTCOMES:
Intensity and longevity of antigen specific T-cell mediated immune responses to the neoantigen vaccine | Up to 12 months
Time to progression | Up to 18 months
Duration of response | Up to 12 months
Clinical benefit rate (minor response or better) | After 6 cycles (168 days)
  Assessed by the modified International Myeloma Working Group criteria for multiple myeloma.
Overall survival | Up to 12 months

OTHER OUTCOMES:
Rate of minimal residual disease negativity at complete remission | Up to 12 months
  Assessed based on bone marrow aspirates.
Molecular and cellular profiling | Up to 12 months
Immunophenotypic analysis | Up to 12 months
  Will assess dendritic, T-, B-, natural killer (NK)- and NKT-cells, and inhibitory/activation markers on tumor cells at baseline (bone marrow and peripheral blood), day 1 of each cycle (peripheral blood only) and at completion of 6 cycles of therapy (bone marrow and peripheral blood) in bone marrow aspirate samples and/or peripheral blood.
Identification of shared human leukocyte antigen class I-restricted antigens that can be targeted with immunotherapy | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Krina Patel, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2023-02-15): https://cdn.clinicaltrials.gov/large-docs/43/NCT03631043/ICF_000.pdf